CLINICAL TRIAL: NCT00606242
Title: A Randomized Double Blind Study of the Dose Response Effects of Fluticasone Propionate on Hypertonic-saline Induced Bronchoconstriction in Asthmatic Subjects
Brief Title: Dose Response Effects of Inhaled Fluticasone on Airway Effects of Hypertonic-saline in Asthma
Acronym: FluSAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); GlaxoSmithKline (Industry)
Responsible Party: John Fahy, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HL6788-15958-08; 5P50HL056385 (NIH)
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose steroid (Active Comparator): Fluticasone, 100 mcg per day
  Interventions: Drug: Fluticasone
- High dose steroid (Active Comparator): Fluticasone, 1000 mcg per day
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Fluticasone — Inhaled Fluticasone, either 100 or 1000 mcg per day
  Other Names: Flovent

SUMMARY:
This study investigates the effect of a inhaled corticosteroid (fluticasone or "Flovent") on airway narrowing induced by hypertonic saline (salty water). The study hypothesis is that fluticasone will be more effective in preventing saline-induced airway narrowing than methacholine-induced narrowing.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma

Exclusion Criteria:

* Habitual cigarette smoking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2000-01; Primary Completion 2002-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
FEV1 | Measured every 2 weeks

SECONDARY OUTCOMES:
PC20 methacholine | Measured every 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States